CLINICAL TRIAL: NCT03197428
Title: Efficacy of Platelet-rich Plasma in the Treatment of Chronic Lateral Ankle Instability
Brief Title: Platelet-rich Plasma for Chronic Lateral Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Superintendent, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA-16026-RD-105066
Record Dates: First submitted 2017-04-13; First posted 2017-06-23 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Ankle Instability; Platelet-rich Plasma
Keywords: Platelet-Rich Plasma; Ankle Injuries; Lateral Ligament, Ankle
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): 15 patients will receive platelet-rich plasma gel applied during the modified Broström-Gould procedure for reconstructing lateral ligament.
  Interventions: Other: Platelet-rich plasma
- Control group (Placebo Comparator): 15 patients will receive whole blood applied during the modified Broström-Gould procedure for reconstructing lateral ligament.
  Interventions: Other: Control

INTERVENTIONS:
Other: Platelet-rich plasma — Platelet-rich plasma gel applied during the modified Broström-Gould procedure for reconstructing lateral ligament
  Arms: PRP group
Other: Control — Whole blood applied during the modified Broström-Gould procedure for reconstructing lateral ligament
  Arms: Control group

SUMMARY:
This study aims to evaluate the effect of platelet-rich plasma (PRP) on chronic lateral ankle instability by comparing the imaging and clinical outcomes between patients receiving PRP and those receiving whole blood during the modified Broström-Gould procedure.

DETAILED DESCRIPTION:
Chronic lateral ankle instability (CAI) in a common foot and ankle problem. It has been linked to recurrent ankle pain, swelling, and even early degenerative change if not properly treated. Lateral ligament reconstruction using modified Broström-Gould procedure is the mainstream in treatment of CAI. Early mobilization is related to better functional outcome, and rapid healing of the repair is the key point to shorten the immobilization time. Platelet-rich plasma (PRP) is a fraction of plasma that contains platelets and multiple growth factors concentrated at high level. Because activated platelets have the potential to release growth factors, PRP has been clinically used to accelerate wound healing and tissue regeneration. However, there is no conclusion regarding the efficacy of PRP on CAI. This clinical trial will investigate the effect of PRP on CAI. Eligible patients will be randomly assigned to receive PRP or whole blood during the modified Broström-Gould procedure. The postoperative imaging and clinical outcomes will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years
* With diagnosis of chronic lateral ankle instability

Exclusion Criteria:

* Poor controlled diabetes
* Peripheral artery obstructive disease
* Skin or soft tissue infection at ankle
* With current or prior history of ankle disease, including degeneration arthritis, fracture, deformity, and cartilage disease.
* With prior history of ankle surgery
* With current or prior history of cancer
* With current or prior history of hematological disease
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
3-month postoperative ankle function evaluated by AOFAS Ankle-Hindfoot score | 3-month postoperative
  Ankle function is evaluated by AOFAS Ankle-Hindfoot score

SECONDARY OUTCOMES:
3-month postoperative ankle pain evaluated by visual analogue scale | 3-month postoperative
  Ankle pain is evaluated by visual analogue scale
3-month postoperative anterior displacement of ankle evaluated by stress radiographs of anterior drawer test | 3-month postoperative
  Anterior displacement is evaluated by the anterior displacement of the talus relative to the tibia on stress radiographs of anterior drawer test.
3-month postoperative lateral tilt of ankle evaluated by stress radiographs of talar tilt test | 3-month postoperative
  Lateral tilt of ankle is evaluated by stress radiographs of talar tilt test.
Percentage of patients with healed ligament evaluated by MRI | 3-month postoperative
  Healing condition of ligament is assessed by MRI.
Percentage of patients with healed ligament evaluated by second look arthroscopy | 3-month postoperative
  Healing condition of ligament is assessed by second look arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No